CLINICAL TRIAL: NCT02919540
Title: Effect of "Kangaroo Mother Care Approach" on Premature Infants' Physiological Outcomes in Jordan
Brief Title: Effect of "Kangaroo Mother Care" on Premature Infants Physiological Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 26/94/2016
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Premature Neonate
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- kangaroo care approach (Experimental): the kangaroo care approach will be implemented for dyads who agree to participate
  Interventions: Other: Kangaroo care approach
- control group (No Intervention): routine care will be implemented

INTERVENTIONS:
Other: Kangaroo care approach — skin to skin contact between stable preterm infants and their naked mother's chest
  Arms: kangaroo care approach

SUMMARY:
This project aims at testing the effect of applying the KMC on the premature infants' physiological outcomes. The findings of this project are expected to contribute to the discipline of preterm infants' care by providing evidence of the benefits, barriers, and facilities of providing the KMC in our Jordanian NICUs.

DETAILED DESCRIPTION:
Premature infants are often unable physiologically to adapt well to the stressful environment of the NICU. These neonates are commonly at risk for the development of short and long term outcomes ranging from mild developmental delay to severe disability. The Kangaroo mother care approach (KMC) is developed to minimize the effect of prematurity and the NICU environmental stressors on premature infants. This project aims at assessing the neonatal nurses' knowledge and attitudes of the application of the KMC approach in the neonatal intensive care unit (NICU), testing the effect of applying the KMC on the premature infants' physiological outcomes, and exploring the mothers' lived experiences of providing KMC for their premature infants. The findings of this project are expected to contribute to the discipline of preterm infants' care by providing evidence of the benefits, barriers, and facilities of providing the KMC in our Jordanian NICUs.

ELIGIBILITY:
Inclusion Criteria:

* all stable preterm or low birth weight infants (stable infants are those who are able to breath unassisted and have no major health problems (WHO, 2003)), weighing more than 1800gm, who are admitted to the NICUs at the time of study and whose mothers consent to participate and willing to practice the KMC with her infant

Exclusion Criteria:

* high risk preterm or low birth weight infants.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02-24 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
Breastfeeding outcome | 4-6 months
  Breastfeeding outcome will be measured for both groups by the numbers of preterm infants discharged on either exclusive or partial breastfeeding

SECONDARY OUTCOMES:
Body temperature | 4-6 months
  Axillary body temperature will be measured using an electronic thermometer
Heart rate (beat per minute) | 4-6 months
  Continuous electrocardiogram (ECG) data will be recorded from two surface chest electrodes
Respiratory activity (breath per minute) | 4-6 months
  A non-invasive signal monitor connected to the infant cardio-respiratory monitor that captures ECG and respiratory data will be used

CONTACTS AND LOCATIONS:
Overall Officials: khulood K. Shattnawi, PhD, Principal Investigator — Jordan University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided